CLINICAL TRIAL: NCT01448811
Title: Impact of Auditory Evoked Potential Index Monitoring on Bronchoscopic Examination in the Mechanical Ventilated Patients - A Prospective, Randomized, Controlled Study
Brief Title: Auditory Evoked Potential Monitoring on Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Chien-Wei Hsu, Assisted Professor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VGHKS96-024
Record Dates: First submitted 2011-10-06; First posted 2011-10-07 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Sedation Method

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- AEP monitoring (Experimental)
  Interventions: Device: AEP monitor
- RSS monitoring (Active Comparator)
  Interventions: Procedure: Ramsay Sedation Scale

INTERVENTIONS:
Device: AEP monitor — In AEP monitoring group, nurses adjusted propofol dose according to AAI values. If AAI>40, titrate up propofol dosage, AAI<25, titrated down propofol dosage.
  Arms: AEP monitoring
Procedure: Ramsay Sedation Scale — During bronchoscopy, nurses adjusted propofol dose according to Ramsay Sedation Scale.
  Arms: RSS monitoring

SUMMARY:
To compare the difference of sedation monitoring for bronchoscopic examination monitoring by auditory evoked potentials (AEP) or Ramsay Sedation Scale (RSS) in mechanical ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients with aged 18 or over and they needed bronchoscopic examination in the ICU were eligible for this study.

Exclusion Criteria:

* patients with pacemaker, neuromuscular blockades, propofol allergy or hearing impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change of mean arterial pressure, heart rate and AAI | 40 minutes
  During bronchoscopy, we recorded AAI number, blood pressure and heart rate every 5 minutes, totally up to 40 minutes.

SECONDARY OUTCOMES:
mean propofol dose use during examination, times of propofol dose adjustment | 40 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Wei Hsu, MD, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung, Taiwan, Taiwan

REFERENCES:
- [Derived] Hsu CW, Sun SF, Chu KA, Lee DL, Wong KF. Monitoring sedation for bronchoscopy in mechanically ventilated patients by using the Ramsay sedation scale versus auditory-evoked potentials. BMC Pulm Med. 2014 Feb 6;14:15. doi: 10.1186/1471-2466-14-15. PMID 24499010